CLINICAL TRIAL: NCT01641081
Title: Phase II, Randomized, Placebo-controlled, Double-blind, Double-dummy, 5-period Complete Crossover Study of the Bronchodilator Effects of Formoterol Fumarate Inhalation Powder in Patients With Mild to Moderate Asthma.
Brief Title: Efficacy and Safety Study to Compare Formoterol Fumerate in the Pressair DPI to the Foradil Aerolizer in Patient With Mild to Moderate Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAC-MD-21
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Results first posted 2016-12-22 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Experimental 1 (Experimental): Formoterol Fumarate in the Pressair Pressair Dry Powder Inhaler (DPI), Low Dose
  Interventions: Drug: Formoterol Fumarate in the Pressair DPI, Low Dose
- Experimental 2 (Experimental): Formoterol fumarate in the Pressair Dry Powder Inhaler (DPI), High Dose
  Interventions: Drug: Formoterol Fumarate in the Pressair DPI, High Dose
- Active Comparator 1 (Active Comparator): Foradil Aerolizer, Low Dose
  Interventions: Drug: Foradil Aerolizer, Low Dose
- Active Comparator 2 (Active Comparator): Foradil Aerolizer, High Dose
  Interventions: Drug: Foradil Aerolizer, High Dose
- Placebo (Placebo Comparator): Dose matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Formoterol Fumarate in the Pressair DPI, Low Dose — Formoterol Fumarate in the Pressair DPI 6 micrograms, twice a day for 14 days
  Arms: Experimental 1
Drug: Formoterol Fumarate in the Pressair DPI, High Dose — Formoterol Fumarate in the Pressair DPI 12 micrograms, twice a day for 14 days
  Arms: Experimental 2
Drug: Foradil Aerolizer, Low Dose — Foradil Aerolizer 12 micrograms, twice a day for 14 days
  Other Names: Formoterol
  Arms: Active Comparator 1
Drug: Foradil Aerolizer, High Dose — Foradil Aerolizer 24 micrograms, twice per day for 14 days
  Other Names: Formoterol
  Arms: Active Comparator 2
Drug: Placebo — Placebo in the Pressair for 14 days
  Arms: Placebo

SUMMARY:
The purpose of this Phase II study is to evaluate efficacy and safety of inhaled formoterol fumarate in the Pressair DPI compared to the Foradil Aerolizer in patients with mild to moderate asthma.

This study will include a screening visit followed by a 4 month treatment period.

ELIGIBILITY:
Inclusions:

* Patients with mild-to-moderate asthma for at least 6 months prior to Visit 1 (as defined in the GINA Guidelines) which is unlikely to exacerbate during the study (e.g., due to seasonal allergen exposure).
* Patients must be on a stable dose of Inhaled Corticosteroids (ICS) for at least 30 days prior to Visit 1. Patients on a combination of ICS/LABA must discontinue the use of LABA and must be on a stable dose of ICS for 30 days prior to Visit 1.
* Qualifying spirometry at Visit 1 demonstrates highest FEV1 is ≤ 85% and ≥ 60% of predicted for age, height, and gender using NHANES III (NHANES 2010) when bronchodilator medications have been withheld the appropriate length of time per the List of Concomitant Medications (Appendix III)
* Patient demonstrates reversibility with an increase in FEV1 of 12% and 200 mL after the administration of 360 µg of albuterol.
* Highest pre-dose FEV1 at Visits 2, 4, 6, 8, and 10 must be within 25% of the qualifying FEV1 at Visit 1

Exclusions:

* Patients with any clinically significant respiratory conditions other than mild to moderate asthma, such as COPD, active tuberculosis, or history of interstitial lung disease
* Patients with a severe asthma exacerbation requiring hospitalization in the previous 12 months
* Patient is not able to withhold use of inhaled short-acting beta-agonist (SABA) for at least 6 hours prior to visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Garcia, MD, Study Director — AstraZeneca
Locations (29):
- United States (29):
  - Forest Investigative Site 909, Phoenix, Arizona
  - Forest Investigative Site 2066, Encinitas, California
  - Forest Investigative Site 1624, Los Angeles, California
  - Forest Investigative Site 1995, Mission Viejo, California
  - Forest Investigative Site 1347, San Jose, California
  - Forest Investigative Site 1996, Centennial, Colorado
  - Forest Investigative Site 1137, Colorado Springs, Colorado
  - Forest Investigative Site 1998, Denver, Colorado
  - Forest Investigative Site 2047, Tampa, Florida
  - Forest Investigative Site 1536, Louisville, Kentucky
  - Forest Investigative Site 1333, Baltimore, Maryland
  - Forest Investigative Site 1431, North Dartmouth, Massachusetts
  - Forest Investigative Site 2041, Minneapolis, Minnesota
  - Forest Investigative Site 1599, St Louis, Missouri
  - Forest Investigative Site 1609, Bellevue, Nebraska
  - Forest Investigative Site 1999, Skillman, New Jersey
  - Forest Investigative Site 1153, Raleigh, North Carolina
  - Forest Investigative Site 1134, Canton, Ohio
  - Forest Investigative Site 1806, Cincinnati, Ohio
  - Forest Investigative Site 1176, Oklahoma City, Oklahoma
  - Forest Investigative Site 2043, Medford, Oregon
  - Forest Investigative Site 1580, Portland, Oregon
  - Forest Investigative Site 2025, Charleston, South Carolina
  - Forest Investigative Site 1155, Dallas, Texas
  - Forest Investigative Site 1332, El Paso, Texas
  - Forest Investigative Site 1370, New Braunfels, Texas
  - Forest Investigative Site 1699, San Antonio, Texas
  - Forest Investigative Site 2011, Seattle, Washington
  - Forest Investigative Site 1997, Madison, Wisconsin

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4059&filename=LAC-MD-21_CSRredacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 29 study centers in the United States
  First patient visit was in June 2012 and last patient visit was in February 2013
Pre-assignment Details: A total of 408 patients were screened; there were 234 screen failures, primarily (225/234) because inclusion/exclusion criteria were not met
Groups:
- Sequence 1: 24 μg Foradil Aerolizer; 12 μg Foradil Aerolizer; Placebo Pressair; Formoterol 12 μg Pressair; Formoterol 6 μg Pressair
- Sequence 2: 12 μg Foradil Aerolizer; Formoterol 12 μg Pressair; 24 μg Foradil Aerolizer; Formoterol 6 μg Pressair; Placebo Pressair
- Sequence 3: Formoterol 12 μg Pressair; Formoterol 6 μg Pressair; 12 μg Foradil Aerolizer; Placebo Pressair; 24 μg Foradil Aerolizer
- Sequence 4: Formoterol 6 μg Pressair; Placebo Pressair; Formoterol 12 μg Pressair; 24 μg Foradil Aerolizer; 12 μg Foradil Aerolizer
- Sequence 5: Placebo Pressair; 24 μg Foradil Aerolizer; Formoterol 6 μg Pressair; 12 μg Foradil Aerolizer; Formoterol 12 μg Pressair
- Sequence 6: Formoterol 6 μg Pressair; Formoterol 12 μg Pressair; Placebo Pressair; 12 μg Foradil Aerolizer; 24 μg Foradil Aerolizer
- Sequence 7: Placebo Pressair; Formoterol 6 μg Pressair; 24 μg Foradil Aerolizer; Formoterol 12 μg Pressair; 12 μg Foradil Aerolizer
- Sequence 8: 24 μg Foradil Aerolizer; Placebo Pressair; 12 μg Foradil Aerolizer; Formoterol 6 μg Pressair; Formoterol 12 μg Pressair
- Sequence 9: 12 μg Foradil Aerolizer; 24 μg Foradil Aerolizer; Formoterol 12 μg Pressair; Placebo Pressair; Formoterol 6 μg Pressair
- Sequence 10: Formoterol 12 μg Pressair; 12 μg Foradil Aerolizer; Formoterol 6 μg Pressair; 24 μg Foradil Aerolizer; Placebo Pressair
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 18 | 18 | 15 | 22 | 17 | 19 | 19 | 17 | 15 | 14
Completed | 17 | 18 | 15 | 22 | 16 | 19 | 18 | 14 | 15 | 14
Not Completed | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 0 | 0
Not completed — Sponsor request (potential unblinding) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 17 | 18 | 15 | 22 | 16 | 19 | 18 | 14 | 15 | 14
Completed | 16 | 18 | 15 | 21 | 16 | 18 | 16 | 14 | 15 | 14
Not Completed | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 16 | 18 | 15 | 21 | 16 | 18 | 16 | 14 | 15 | 14
Completed | 16 | 18 | 14 | 21 | 16 | 18 | 16 | 14 | 14 | 14
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 4
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 16 | 18 | 14 | 21 | 16 | 18 | 16 | 14 | 14 | 14
Completed | 16 | 17 | 14 | 20 | 16 | 18 | 16 | 14 | 14 | 14
Not Completed | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Sequence 7 | Sequence 8 | Sequence 9 | Sequence 10
Started | 16 | 17 | 14 | 20 | 16 | 18 | 16 | 14 | 14 | 14
Completed | 16 | 17 | 12 | 20 | 16 | 18 | 16 | 14 | 14 | 14
Not Completed | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: All patients participating in the crossover study
Arm/Group | Overall Study Population
Number analyzed (Participants) | 174
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.4 (13.2)
Gender [Count of Participants; unit: Participants]
  Female | 91
  Male | 83

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Normalized Forced Expiratory Volume in One Second (FEV1) AUC0-6 After the Morning Dose (Day 14)
Description: AUC0-6 is area under the curve from time 0 to 6 hours Serial spirometry was performed at -60 min predose, at 5 (+5) and 30 (±5) min post-dose, and at 1, 2, 3, 4, and 6 hrs post-dose (±15 min) Change from baseline was baseline of each treatment period The normalized FEV1 AUC0-6 was calculated by means of the trapezoidal method, dividing the area under the curve by the corresponding time intervals
Time Frame: Baseline and up to 6 hrs post-dose (±15 min) on Day 14 of treatment
Population: Intent to treat (ITT) Population defined as all patients in the Safety Population who had a baseline and at least 1 post-baseline FEV1 assessment
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Foradil 24 μg; Foradil 12 μg: Administered via Aerolizer
- Formoterol 12 μg; Formoterol 6 μg; Placebo: Administered via Pressair
Arm/Group | Foradil 24 μg | Foradil 12 μg | Formoterol 12 μg | Formoterol 6 μg | Placebo
Number analyzed (Participants) | 155 | 151 | 155 | 159 | 154
Liters | 0.3196 (0.0382) | 0.3076 (0.0382) | 0.2795 (0.0382) | 0.2726 (0.0381) | 0.0552 (0.0382)
Statistical Analysis 1: Comparison: Foradil 24 μg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment and period as fixed effects, and baseline FEV1 values at each period as a covariate; Least squares mean difference = 0.2644, 95% CI 2-sided [0.2353 to 0.2934], Standard Error of Mean 0.0148
Statistical Analysis 2: Comparison: Foradil 12 μg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment and period as fixed effects, and baseline FEV1 values at each period as a covariate; Least squares mean difference = 0.2524, 95% CI 2-sided [0.2218 to 0.2830], Standard Error of Mean 0.0156
Statistical Analysis 3: Comparison: Formoterol 12 μg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment and period as fixed effects, and baseline FEV1 values at each period as a covariate; Least squares mean difference = 0.2242, 95% CI 2-sided [0.1941 to 0.2544], Standard Error of Mean 0.0153
Statistical Analysis 4: Comparison: Formoterol 6 μg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Treatment and period as fixed effects, and baseline FEV1 values at each period as a covariate; Least squares mean difference = 0.2174, 95% CI 2-sided [0.1887 to 0.2461], Standard Error of Mean 0.0146

2. Secondary Outcome: Change From Baseline in Normalized FEV1 AUC0-6 After the Morning Dose (Day 1)
Description: AUC0-6 is area under the curve from time 0 to 6 hours Serial spirometry was performed at -60 min predose, at 5 (+5) and 30 (±5) min post-dose, and at 1, 2, 3, 4, and 6 hrs post-dose (±15 min) Change from baseline was baseline of Period 1 The time-normalized FEV1 AUC0-6 was calculated by means of the trapezoidal method, dividing the area under the curve by the corresponding time intervals
Time Frame: Baseline and up to 6 hrs post-dose (±15 min) on Day 1 of treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Foradil 24 μg | Foradil 12 μg | Formoterol 12 μg | Formoterol 6 μg | Placebo
Number analyzed (Participants) | 163 | 155 | 159 | 158 | 154
Liters | 0.3544 (0.0196) | 0.3068 (0.0198) | 0.2712 (0.0197) | 0.2204 (0.0197) | 0.0306 (0.0198)

ADVERSE EVENTS:
Time Frame: Day 14±1 of the final treatment period (Period 5)
Description: The Safety Population consisted of all patients screened, randomized to a treatment sequence, and who took at least one dose of double-blind investigational product The total number of patients in the Safety Population was 174; due to study drop-out and the crossover study design, not all patients received all treatments
Arm/Group | Foradil 24 μg | Foradil 12 μg | Formoterol 12 μg | Formoterol 6 μg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/167 | 2/163 | 0/164 | 0/166 | 0/165
Other Adverse Events (participants affected / at risk) | 10/167 | 2/163 | 2/164 | 1/166 | 0/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Foradil 24 μg (N=167) | Foradil 12 μg (N=163) | Formoterol 12 μg (N=164) | Formoterol 6 μg (N=166) | Placebo (N=165)
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Foradil 24 μg (N=167) | Foradil 12 μg (N=163) | Formoterol 12 μg (N=164) | Formoterol 6 μg (N=166) | Placebo (N=165)
Tremor (Nervous system disorders) | 10 | 2 | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results by the PI will be subject to mutual agreement between the PI and sponsor.